CLINICAL TRIAL: NCT00361283
Title: Systemic Immunomodulatory Effects and Pharmacogenetics of Atorvastatin in Early Atherosclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Heart Association (Other); American College of Clinical Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0435278B
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-04

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- atorvastatin (Other): 80mg of atorvastatin given once daily for 16 weeks
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — atorvastatin 80mg tablets given by mouth once daily for 16 weeks with follow-up visits every 4 weeks
  Other Names: Lipitor

SUMMARY:
The purpose of the study is to test whether atorvastatin (also known as Lipitor) has anti-inflammatory effects in people with no known heart disease or high cholesterol. We also are investigating whether or not genetic differences between people plays a role in the drug response.

DETAILED DESCRIPTION:
All subjects received 16 weeks of Atorvastatin after a two week run in. Key dependent variables were the 16 week value minus the baseline value (post run-in). Last observation carried forward was used for missing values. The key comparisons are for two groups OATP1B1 reduced carriers and on-carriers and their association with Cytokines and Lipids. Secondarily, we were interested in changes over the 16 weeks for the pooled sample, irrespective of genetics.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Normocholesterolemic

Exclusion Criteria:

* Cardiovascular disease or risk equivalents
* Malignancy
* Active alcohol abuse
* Contraindications to statins
* Interacting drugs
* Chronic anti-inflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-06; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Frye, PharmD, PhD, Principal Investigator — University of Florida College of Pharmacy
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University of Florida Clinical Research Center. Study started June 2004 and ended January 9, 2009.
Period: Overall Study
Arm/Group | Atorvastatin
Started | 108
Completed | 81
Not Completed | 27
Not completed — Lost to Follow-up | 27

BASELINE CHARACTERISTICS:
Arm/Group | Atorvastatin
Number analyzed (Participants) | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 107
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 31.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 108

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Level: Week 16-baseline in Ena-78
Description: We take difference week 16 minus week 0 for ENA-78 and use a one sample t comparison.
Time Frame: 16 weeks after baseline
Population: Power calculation
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Atorvastatin 80 MG/Day: Atorvastatin 80 MG/day
Arm/Group | Atorvastatin 80 MG/Day
Number analyzed (Participants) | 81
pg/ml | -111.2 (690.5)
Statistical Analysis 1: Comparison: Atorvastatin 80 MG/Day; The study in healthy volunteers was to compare levels at baseline to 16 weeks in ENA-78, a cytokine. The one sample t-test was used to obtain the result; Test type: Superiority or Other; p = 0.15, t-test, 2 sided — No confounders were controlled for as each person is his/her own control; Mean Difference (Net) = -111, 95% CI 2-sided [-264 to 42], Standard Error of Mean 76.7

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 14/108
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=108)
Muscle aches (Musculoskeletal and connective tissue disorders) | 14 (14)
Headache (General disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No